CLINICAL TRIAL: NCT00702039
Title: Effect of Music Therapy on Patients Undergoing Intravitreal Injections
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 0702002303
Record Dates: First submitted 2008-04-01; First posted 2008-06-19 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Intravitreal Injections; Patient Satisfaction; Patient Anxiety
MeSH Terms: conditions — Patient Satisfaction | interventions — Music Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Those patients receiving intravitreal injections who will be listening to classical music during injection.
  Interventions: Other: Music Therapy
- 2: Those patients receiving intravitreal injections who will not be listening to any music during injection.
  Interventions: Other: No Music

INTERVENTIONS:
Other: No Music — No music will be played in patients in arm 2 of the study.
  Groups: 2
Other: Music Therapy — Classical music being played during intravitreal injection.
  Groups: 1

SUMMARY:
Multiple studies in various specialties, including ophthalmology, are reported in the literature that show that playing music during a procedure (dubbed music therapy) increases patient satisfaction and may reduce patient anxiety and stress levels.

There is no study in the literature that assesses the effects of listening to music in patients undergoing intravitreal injections. This study aims to assess whether listening to music improves patient satisfaction or reduces their anxiety levels in subjects undergoing intravitreal injections.

ELIGIBILITY:
Inclusion Criteria:

* Those patients at least 18 years old already scheduled for intravitreal injections.

Exclusion Criteria:

* Those patients not interested in participating in the study or not capable of filling out the questionnaire secondary to limited mental capability.
* Non- English speaking subjects will be excluded from the study.
* Those patients that participated in the study will not be allowed to participate a second time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving intravitreal injections seen at the Yale Eye Center.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-02; Primary Completion 2009-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
This study aims to assess what affects music therapy has on patients receiving intravitreal injections. The subject will take a Satisfaction Survey after the procedure and an Anxiety Survey before and after the injection. | Before and after the subject's intravitreal injection.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Adelman, MD, Principal Investigator — Yale University Department of Ophthalmology
Locations (1):
- Yale Eye Center, New Haven, Connecticut, United States